CLINICAL TRIAL: NCT01269905
Title: Choice of Valve Substitute in the Era of Oral Anticoagulation Self-Management
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Other Study IDs: COAG-001
Record Dates: First submitted 2011-01-03; First posted 2011-01-04 (Estimated); Last update posted 2011-01-04 (Estimated); Status verified 2005-01

CONDITIONS: Anticoagulation; Mechanical Heart Valve Replacement

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- Group A: Group A patients received mechanical heart valve replacement MHVR (and were educated in INR self-management using the Coagu-Check monitor.
- Group B: Group B patients received MHVR and their anticoagulation was managed by their general practitioners.
- Group C: Group C patients received stentless bioprosthesis, with initial 6 weeks on oral anticoagulation managed by their general practitioners.

SUMMARY:
The optimal valve substitute for patients between 60-70 years is controversial. We compared anticoagulation-related adverse events (ARAE) in patients receiving mechanical heart valve replacement (MHVR) on INR self-management vs. stentless bioprosthesis, to assess whether the risk of structural valve deterioration (SVD) is still out-weighted by the benefit of not requiring permanent anticoagulation.

ELIGIBILITY:
Inclusion Criteria:

* heart valve replacement

Exclusion Criteria:

* CABG
* Afib

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients received heart valve replacement and were retrospectively allocated in three groups
Sampling Method: Non-Probability Sample